CLINICAL TRIAL: NCT03638024
Title: Predictive Value of Cell-free Fetal DNA Concentration in the Maternal Plasma for Abnormal Placental Invasion in Cases of Placenta Previa.
Brief Title: Cell-free Fetal DNA Concentration in Cases of Abnormal Placental Invasion .
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr- dina yahia mansour, Lecturer of Obstetrics and Gynecology Ain Shams University, Ain Shams Maternity Hospital
Other Study IDs: Cell free fetal DNA
Record Dates: First submitted 2018-05-09; First posted 2018-08-20 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Placenta Accreta; Placenta Percreta; Placenta Increta; Placenta Previa
MeSH Terms: conditions — Placenta Accreta; Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Maternal plasma cell free fetal DNA levels will be measured in 25 women with one or more previous cesarean section and placenta previa anterior only or with ultrasound finding suggestive of placental adhesion or invasion (accreta , increta or percreta).
  Interventions: Diagnostic Test: Maternal plasma cell free fetal DNA levels
- Control group: Maternal plasma cell free fetal DNA levels will be measured in 25 matched control with normally situated placenta without ultrasound finding suggestive of placental adhesion or invasion.
  Interventions: Diagnostic Test: Maternal plasma cell free fetal DNA levels

INTERVENTIONS:
Diagnostic Test: Maternal plasma cell free fetal DNA levels — Measurement Maternal plasma cell free fetal DNA levels in both groups (study and control groups)

SUMMARY:
Cell free fetal DNA might predict abnormal placental invasion

DETAILED DESCRIPTION:
This study aims to evaluate whether measurement of cell-free fetal DNA in the maternal plasma can be predictive of abnormal invasion in cases of placenta previa.

ELIGIBILITY:
Inclusion criteria:

1. Maternal age range from 20-40 years old.
2. Parity: para 1- para 5.
3. Body mass index range from 18-25 kg/m2.
4. Singleton pregnancy carrying male fetuses.
5. Gestational age range from 28-34 weeks.

Exclusion criteria:

1. Multifetal pregnancy.
2. Hypertension, preterm labor and intrauterine growth restriction.
3. Patients taking a tocolytic agent or those with uterine bleeding at or after blood sampling.

   * Since these complications may increase the level of cell-free fetal DNA.
4. Accidental hemorrhage.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Study group (1): 25 women with one or more previous cesarean section and placenta previa anterior only or with ultrasound finding suggestive of placental adhesion or invasion (accreta , increta or percreta).
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-03-03 (Estimated); Study Completion 2019-04-03 (Estimated)

PRIMARY OUTCOMES:
Predictive value of maternal plasma cell free DNA | 4 months
  Prediction of abnormal placental invasion in cases of placenta previa.
  Primary aim: Is to evaluate whether measurement of cell-free fetal DNA in the maternal plasma can be predictive of abnormal placental invasion in cases of placenta previa.
  Secondary aim: To decrease maternal morbidity and mortality by early prenatal diagnosis of abnormal placental invasion in placenta previa

SECONDARY OUTCOMES:
maternal morbidity | 4 months
  maternal morbidity

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Maternity Hospital, Cairo, Egypt